CLINICAL TRIAL: NCT05251428
Title: A Randomized Control Trial to Evaluate Incision Versus Excision of A1 Pulley for Trigger Finger
Brief Title: Trigger Finger Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Eric Wagner, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003754
Record Dates: First submitted 2022-02-01; First posted 2022-02-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- excision of the A1 pulley (Experimental)
  Interventions: Procedure: Excision of the A1 pulley
- incision of the A1 pulley in the standard fashion (Active Comparator)
  Interventions: Procedure: Incision of the A1 pulley in the standard fashion

INTERVENTIONS:
Procedure: Excision of the A1 pulley — Participants will undergo excision of the A1 pulley. Wounds will then be irrigated and closed in the standard fashion.
  Other Names: Intervention Group
  Arms: excision of the A1 pulley
Procedure: Incision of the A1 pulley in the standard fashion — Participants will undergo incision of the A1 pulley in the standard fashion. Wounds will then be irrigated and closed in the standard fashion.
  Other Names: Standard of care group
  Arms: incision of the A1 pulley in the standard fashion

SUMMARY:
Trigger finger is a common condition of the hand caused by the thickening of the A1 pulley or flexor tendon that alters the way in which the flexor tendon glides within the tendon sheath.

The purpose of this study is to evaluate the efficacy of excision versus incision of the A1 pulley for the trigger finger. Researchers hypothesize that excision of the A1 pulley would result in lower trigger finger recurrence rates, better pain relief, reduced soreness & stiffness as well as higher final Patient-Reported Outcomes Measurement (PROMs).

This will be investigated via a randomized controlled study involving patients randomized in either of the aforementioned surgical treatment groups, which are both standards of care, at the Musculoskeletal Institute or at the Emory University Orthopaedic and Spine Hospital. Patients will then follow up in the clinic at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year to assess their outcomes measures stated in the protocol document. All work related to this project will take place at the Emory Sports Medicine Complex, Emory Executive Park, Emory Musculoskeletal Institute, and the Emory University Orthopaedic and Spine Hospital. Patients will not be compensated for participating in this study. Patients who are undergoing trigger finger surgery will be identified by their Orthopaedic surgeon who is a member of the study team. The surgeon will briefly discuss participation with the patient and make clear study expectations.

DETAILED DESCRIPTION:
Trigger finger is a common condition of the hand that affects up to 2.6% of the adult population over the course of their lifetimes. This prevalence is even higher in patients with diabetes affecting 5-20% of people. The condition is caused by the thickening of the A1 pulley or flexor tendon that alters the way in which the flexor tendon glides within the tendon sheath. While first-line therapy for this condition is conservative treatment through activity modification, bracing, and corticosteroid injections, this fails a reported 20-50% of the time. In cases in which conservative management failure occurs, surgery is the next line of treatment. The purpose of this study is to evaluate the efficacy of excision versus incision of the A1 pulley for the trigger finger. The research team hypothesizes that excision of the A1 pulley would result in lower trigger finger recurrence rates, better pain relief, reduced soreness & stiffness as well as higher final PROMs.

Surgery can be performed either percutaneously or open. Rates of persistent triggering in the percutaneous release group range from 7 to 9%. Additionally, even with open procedures, there is some risk of persistent triggering or symptom recurrence. A study by Everding et al. reported a recurrent triggering rate of 2.6% in their cohort of 795 patients who underwent open trigger finger release. A review of 209,634 patients who underwent trigger digit release from the PearlDiver Database reported a revision rate of 0.4% at 1 year and 0.64% at 3 years. Finally, a retrospective study by Bruijnzeel et al. demonstrated a 0.6% risk of persistent triggering and a 0.3% risk of recurrence in their sample of 1,598 patients. Risk factors for revision include Dupuytren's disease, rheumatoid arthritis, liver, disease, obesity, tobacco use, peripheral vascular disease, diabetes mellitus, and age under 65 years. In cases of recurrence, the procedure can be repeated to release any remaining portion of the A1 pulley, partial release of the A2, or release of the ulnar slip of flexor digitorum superficialis. Two biomechanical studies have demonstrated that the entire A1 pulley and up to 50% of the A2 pulley can be released with minimal risk for bowstringing.

There have also been studies assessing the use of different incision types for open procedures and their effects on scar formation. Kazmers et al. compared scar formation from trigger finger release through a transverse skin incision versus a longitudinal incision and found no difference in DASH scores, complication rates, or scar quality metrics in the 61 patients studied. Additionally, a study comparing a transverse incision at the distal palmar crease, a transverse incision 2-3 mm distal to the distal palmar crease, and a longitudinal incision at the level of the A1 pulley demonstrated similar results between the longitudinal incision and the incision 2-3 mm distal to the distal palmar crease with no difference in scar volume as measured by ultrasound. There have been no studies to date assessing the effect of complete A1 pulley resection in comparison to longitudinal release of the A1 pulley. Theoretically, resection of the A1 pulley should reduce the rate of persistent triggering and recurrence and thus result in superior patient outcomes; however, this has yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* All patients undergoing surgery for trigger finger syndrome
* Patients willing and able to provide informed consent

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Change in the pain score | Baseline and 6 weeks
  Participants will be asked to complete questionnaires to evaluate their pain at each follow-up visit. The Visual Analog Scale will be the subjective measurement to evaluate changes in pain scores, with values ranging from 0 (no pain) to 10 (very severe pain). A higher score indicates worse pain.

OTHER OUTCOMES:
Change in the range of motion (ROM) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, and 1 year
  Participants will be asked to complete questionnaires to evaluate their stiffness at each follow-up visit. The range of motion (ROM) will be measured using a finger goniometer ranging from 0 to 180 degrees. Additional hand function outcomes will be measured using the Disabilities of Arm, Shoulder, and Hand Questionnaire (DASH) which consists of subjectively rating the difficulty of a list of activities of daily living from 0-5 (0: no difficulty, 5=unable).
Change in patients' reported Working status | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, and 1 year
  The Upper Extremity Patient-Reported Outcomes Program (PROM) is a patient outcomes questionnaire that will be completed by the study participant at every visit. This questionnaire is administered electronically on a Microsoft tablet in the study room with the study participants' own password-secured profile log. The questionnaire consists of the subjective scores described above (DASH, VAS) as well as questions pertaining to current work status (unable to work, employed, caregiver/homemaker, retired).
Change in the pain score | Baseline, 2 weeks, 3 months, 6 months, and 1 year
  Participants will be asked to complete questionnaires to evaluate their pain at each follow-up visit. The Visual Analog Scale will be the subjective measurement to evaluate changes in pain scores, with values ranging from 0 (no pain) to 10 (very severe pain). A higher score indicates worse pain.
Recurrent trigger finger after A1 pulley release | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, and 1 year
  The research team will assess participants for recurrence of their symptoms. Recurrence of the trigger finger is defined as finger triggering after the surgery. Finger triggering is described as the involved finger becoming stuck in a bent position and straightening with a snap, like a trigger being pulled and released. This is a clinical manifestation of the pathology, evaluated and determined by the treating surgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wagner, MD, MS, Principal Investigator — Emory University
Locations (6):
- United States (6):
  - Emory Orthopedic and Spine Hospital, Atlanta, Georgia
  - 12 Executive Park Drive, Atlanta, Georgia
  - Emory Musculoskeletal Institute, Atlanta, Georgia
  - Emory Orthopaedics and Spine Center, Atlanta, Georgia
  - Emory at Dunwoody, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No